CLINICAL TRIAL: NCT01816295
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel Study With an Open-Label Extension to Assess the Impact of Testosterone Solution on Total Testosterone, Sex Drive and Energy in Hypogonadal Men
Brief Title: A Study in Men With Low Testosterone to Measure the Effects of Testosterone Solution on Testosterone Levels, Sex Drive and Energy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14396; I5E-MC-TSAT (Other: Eli Lilly and Company); 2012-004866-16 (EudraCT Number)
Record Dates: First submitted 2013-03-19; First posted 2013-03-22 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-11

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone Propionate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Solution (Placebo Comparator): Placebo Solution applied topically once daily for 12 weeks.
  Interventions: Drug: Placebo Solution
- Testosterone Solution (Experimental): Testosterone Solution 60 milligram (mg) applied topically once daily with possible titration down to 30 milligram per day (mg/day) or up to 120 mg/day for 12 weeks and optional extension for 24 weeks.
  Interventions: Drug: Testosterone Solution

INTERVENTIONS:
Drug: Testosterone Solution — Administered topically to axillae.
  Other Names: Axiron; Testosterone Solution 2%; LY900011
  Arms: Testosterone Solution
Drug: Placebo Solution — Administered topically to axillae.
  Arms: Placebo Solution

SUMMARY:
The main purpose of this study is to evaluate if testosterone solution can raise testosterone hormone levels into the normal range, and also improve levels of sexual arousal, interest and drive and/or energy level, in men with low testosterone and decreased sexual arousal, interest and drive and/or decreased energy. The study will last about 16 weeks, followed by an optional 24 week open label treatment phase to investigate the long term safety of testosterone solution.

ELIGIBILITY:
Inclusion Criteria:

* Total testosterone level <300 nanogram per deciliter (ng/dL) [10.4 nanomole per Liter (nmol/L)] at each of 2 screening visits
* At least 1 symptom of testosterone deficiency, which must include decreased energy or decreased sexual drive
* Prostate Specific Antigen (PSA) <4 nanogram per milliliter (ng/ml) at screening

Exclusion Criteria:

* Sexual partner who is or becomes pregnant at any time during the study
* Use of long-acting intramuscular (IM) testosterone undecanoate or testosterone pellets in the 6-month period prior to screening
* Body Mass Index (BMI) >37 kilogram per square meter (kg/m^2) at screening
* Severe lower urinary tract symptoms and/or significant prostate enlargement
* Prolactin lab test result of >30 ng/mL at screening
* Hemoglobin A1c (HbA1c) >11% at screening
* Hematocrit ≥50% (>54% at elevated altitude) at screening
* Current use of any medications, herbal, and/or nutritional supplements that can interfere with testosterone
* Dermatologic condition in underarm area that might interfere with testosterone absorption (for example, eczema) or be exacerbated by topical testosterone replacement therapy
* Currently receiving treatment with cancer chemotherapy or antiandrogens
* Chronic use of systemic glucocorticoids (use for >14 days within the 3 months prior to screening); use of non-testosterone anabolic steroids within 12 months prior to screening
* Competitive athletes involved in a sport in which they may be screened for anabolic steroids
* History of use of estrogenizing agents within 12 months prior to screening
* History of luteinizing hormone-releasing hormone antagonist or agonist treatment in the last 6 months prior to screening
* History of clomiphene or other anti-estrogen treatment in the 3 months prior to screening
* Use of finasteride within 3 months prior to screening, or use of dutasteride within 6 months prior to screening
* Current use of warfarin or phenprocoumon
* History of frequent opioid use: >1 time/week during any week within 30 days prior to screening
* Current use of dopamine receptor agonists (cabergoline, pergolide, bromocriptine)
* Have a history of significant central nervous system injuries or disease (including stroke, spinal cord injury, or multiple sclerosis) within 6 months prior to screening
* Systolic blood pressure >170 or <90 millimeter of mercury (mm Hg) or diastolic blood pressure >100 or <50 mm Hg at screening or a history of malignant hypertension
* History of unstable angina as defined by Braunwald Classification of Unstable Angina or angina occurring during sexual intercourse in the last 6 months
* History of any of the following coronary conditions within 90 days of screening: myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention (angioplasty or stent placement)
* Have any supraventricular arrhythmia with an uncontrolled ventricular response [mean heart rate >100 beats per minute (bpm)] at rest, or have any history of spontaneous or induced sustained ventricular tachycardia (heart rate >100 bpm for ≥30 seconds), or use of an automatic internal cardioverter-defibrillator
* Have a history of sudden cardiac arrest
* Exhibit any evidence of congestive heart failure [New York Heart Association (NYHA) Class 2 or above], within 6 months prior to screening
* Have had a new, significant cardiac conduction defect within 90 days prior to screening
* Clinical suspicion (or history) of prostate cancer during digital rectal examination at screening
* Known or suspected breast cancer (or history of breast cancer) or other active cancer (with the exception of nonmelanotic skin cancer)
* Exhibit evidence of severe renal impairment [creatinine clearance <30 milliliter per minute (mL/min) as determined by the Cockcroft-Gault formula] at screening
* Exhibit a history of severe liver disease or clinical evidence of hepatic impairment at screening
* Have a history of human immunodeficiency virus (HIV) infection
* Severe sleep apnea
* Untreated hypothyroidism, hypercortisolism or other significant endocrinopathy (other than hypogonadism) that contributes to symptoms of low energy or fatigue

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (85):
- United States (45):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homewood, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chandler, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tempe, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oviedo, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crystal Lake, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbelt, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Englewood, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bala-Cynwyd, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mt. Pleasant, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingsport, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clinton, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
- Canada (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barrie, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hettstedt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holzminden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
- Italy (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ancona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rozzano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- South Korea (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeonju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pusan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aravaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coslada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Majadahonda
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hathersage Road, Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barnsley

REFERENCES:
- [Derived] Lee H, Hwang EC, Oh CK, Lee S, Yu HS, Lim JS, Kim HW, Walsh T, Kim MH, Jung JH, Dahm P. Testosterone replacement in men with sexual dysfunction. Cochrane Database Syst Rev. 2024 Jan 15;1(1):CD013071. doi: 10.1002/14651858.CD013071.pub2. PMID 38224135
- [Derived] Brock G, Heiselman D, Maggi M, Kim SW, Rodriguez Vallejo JM, Behre HM, McGettigan J, Dowsett SA, Hayes RP, Knorr J, Ni X, Kinchen K. Effect of Testosterone Solution 2% on Testosterone Concentration, Sex Drive and Energy in Hypogonadal Men: Results of a Placebo Controlled Study. J Urol. 2016 Mar;195(3):699-705. doi: 10.1016/j.juro.2015.10.083. Epub 2015 Oct 20. PMID 26498057

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Solution: Placebo solution applied topically to axillae once daily for 12 week double-blind treatment period. In optional open label extension (OLE) period, 60 milligram (mg) testosterone solution applied topically to axillae once daily with possible down/up titration (30 - 120 mg/day) for 24 weeks.
- Testosterone Solution: Sixty mg testosterone solution applied topically to axillae once daily with possible down/up titration (30 - 120 mg/day) for 12 week double-blind treatment period. Optional OLE period starting at 60 mg/day with possible down/up titration (30 - 120 mg/day) for 24 weeks.
Period: Double Blind Phase
Arm/Group | Placebo Solution | Testosterone Solution
Started | 357 | 358
Received Study Drug | 356 | 354
Completed | 294 | 302
Not Completed | 63 | 56
Not completed — Adverse Event | 11 | 8
Not completed — Entry Criteria Not Met | 0 | 2
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 2 | 2
Not completed — Protocol Violation | 17 | 11
Not completed — Sponsor Decision | 8 | 8
Not completed — Withdrawal by Subject | 22 | 20
Period: OLE Phase
Arm/Group | Placebo Solution | Testosterone Solution
Started | 275 (Participants who completed the DBP and still met eligibility criteria had option to enroll in OLE.) | 283 (Participants who completed the DBP and still met eligibility criteria had option to enroll in OLE.)
Completed | 222 | 227
Not Completed | 53 | 56
Not completed — Adverse Event | 17 | 15
Not completed — Death | 1 | 0
Not completed — Entry Criteria Not Met | 3 | 5
Not completed — Lost to Follow-up | 5 | 5
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 4 | 4
Not completed — Sponsor Decision | 7 | 9
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Lack of Efficacy | 3 | 7

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Solution | Testosterone Solution | Total
Number analyzed (Participants) | 357 | 358 | 715
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.35) | 54.7 (10.58) | 55.3 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 357 | 358 | 715
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 57 | 108
  Not Hispanic or Latino | 280 | 279 | 559
  Unknown or Not Reported | 26 | 22 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 38 | 45 | 83
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 26 | 24 | 50
  White | 282 | 281 | 563
  More than one race | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  East Asia | 34 | 40 | 74
  Europe | 63 | 57 | 120
  South America | 28 | 30 | 58
  North America | 232 | 231 | 463
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m²)] — BMI is an estimate of body fat based on body weight divided by height squared.
  kilogram per square meter (kg/m²) | 30.9 (4.21) | 30.3 (4.06) | 30.6 (4.14)
Symptoms of Hypogonadism [Number; unit: participants]
  Only Low Energy | 49 | 47 | 96
  Only Decreased Sexual Drive | 39 | 40 | 79
  Both Symptoms Present | 269 | 271 | 540

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Serum Testosterone Concentration Within Normal Range at Week 12
Description: Normal range for total serum testosterone was defined as 300 to 1050 nanograms per deciliter (ng/dL).
Time Frame: Week 12
Population: All randomized participants who completed 12 weeks of treatment and had non-missing testosterone concentration at week 12.
Measure: Number; unit: participants
Arm/Group | Placebo Solution | Testosterone Solution
Number analyzed (Participants) | 287 | 297
participants | 43 | 217
Statistical Analysis 1: Comparison: Placebo Solution vs Testosterone Solution; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: Change From Baseline to Week 12 in Sexual Arousal, Interest, and Drive (SAID) Scale Scores
Description: The SAID Scale is a self-administered instrument used to assess sexual arousal, interest, and sex drive in men with symptomatic hypogonadism. The SAID consists of 5 questions that were scored on a scale from 1 to 5, with "5" corresponding to greater levels of sexual arousal, interest, or drive. The SAID Scale total score was computed by summing the item scores and linearly transforming the sum to a 0 to 100 scale, with higher scores corresponding to greater sexual arousal, interest, and drive. Least squares (LS) mean change from baseline was calculated using an analysis of covariance (ANCOVA) with treatment group and the baseline value as covariates.
Time Frame: Baseline, Week 12
Population: Randomized participants who reported low sex drive at baseline with non-missing SAID Scale data at baseline and at least one post baseline visit. Missing data endpoints were imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Solution | Testosterone Solution
Number analyzed (Participants) | 257 | 244
units on a scale | 6.3 (0.99) | 11.4 (1.02)
Statistical Analysis 1: Comparison: Placebo Solution vs Testosterone Solution; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 5.1, 99.5% CI 2-sided [1.05 to 9.07], Standard Error of Mean 1.42

3. Secondary Outcome: Change From Baseline to Week 12 in Hypogonadism Energy Diary (HED) Scores
Description: The HED is a self-administered instrument used to assess real-time energy levels in men with symptomatic hypogonadism. It consists of 2 questions that were scored on a scale from 0 to 10, with "10" corresponding to "Full of Energy" or "Not Tired at All" (The Tiredness scale was reverse-mapped, as it was collected with "10" corresponding to "Extreme Tiredness"). The questionnaire was completed 3 times daily (forming 6 unique items) for 7 consecutive days. Item scores were computed by averaging the values for each item across 7 days. If more than 2 days were missing for an item, the item score was missing. The total score was computed by summing the item scores and linearly transforming the sum to a 0 to 100 scale, with higher scores corresponding to greater energy. If any item score was missing, the total score was missing. LS mean change from baseline was calculated using ANCOVA with treatment group and the baseline value as covariates.
Time Frame: Baseline, Week 12
Population: Randomized participants who reported low energy at baseline with non-missing HED questionnaire at baseline and at least one post baseline visit. Missing data endpoints were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Solution | Testosterone Solution
Number analyzed (Participants) | 243 | 230
units on a scale | 7.5 (0.87) | 10.5 (0.89)
Statistical Analysis 1: Comparison: Placebo Solution vs Testosterone Solution; Test type: Superiority or Other; p = 0.019, ANCOVA; Mean Difference (Net) = 2.9, 99.5% CI 2-sided [-0.59 to 6.45], Standard Error of Mean 1.25

4. Other Pre Specified Outcome: Change From Baseline in Total International Prostate Symptom Score (IPSS)
Description: The IPSS is a self-administered instrument used to assess for the severity of lower urinary tract symptoms. The IPSS consists of 7 questions that were scored on a scale from 0 (none/no symptoms) to 5 (frequent symptoms), for a total score range of 0 to 35. Higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. LS mean change from baseline was calculated using ANCOVA with treatment group and the baseline value as covariates.
Time Frame: Baseline, Week 12, Week 36
Population: All randomized participants with non-missing baseline IPSS measurement and at least one non-missing post baseline IPSS measurement. Missing data endpoints were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Solution | Testosterone Solution
Number analyzed (Participants) | 320 | 324
units on a scale
  Change from Baseline to Week 12 | -0.7 (0.24) | -0.9 (0.24)
  Change from Baseline to Week 36 (n=247, 255) | -0.7 (0.28) | -0.7 (0.27)
Statistical Analysis 1: Comparison: Placebo Solution vs Testosterone Solution; Change from Baseline to Week 12; Test type: Superiority or Other; p = 0.442, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.94 to 0.41], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Placebo Solution vs Testosterone Solution; Change from Baseline to Week 36; Test type: Superiority or Other; p = 0.905, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.82 to 0.72], Standard Error of Mean 0.39

5. Secondary Outcome: Number of Participants With Prostate Specific Antigen (PSA) >4 Nanogram/Milliliter (ng/mL)
Time Frame: Double Blind Baseline, Week 12, Open Label Baseline, Week 36
Population: All participants with non-missing PSA result at the specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo Solution | Testosterone Solution
Number analyzed (Participants) | 350 | 347
participants
  Double-Blind Baseline (n=350, 347) | 1 | 0
  Week 12 (n=289, 299) | 3 | 4
  Open Label Baseline (n=269, 278) | 0 | 0
  Week 36 (n=219, 223) | 4 | 4

ADVERSE EVENTS:
Description: Analysis population includes all evaluable, randomized patients who received at least one dose of study drug.
Groups:
- Placebo Solution - Double Blind: Placebo solution applied topically to axillae once daily for 12 week double-blind treatment period.
- Testosterone Solution - Double Blind: Sixty mg testosterone solution applied topically to axillae once daily with possible down/up titration (30 - 120 mg/day) for 12 week double-blind treatment period.
- Testosterone Solution - OLE: Sixty mg testosterone solution applied topically to axillae once daily at 60 mg/day with possible down/up titration (30 - 120 mg/day) for 24 weeks in optional OLE period.
Arm/Group | Placebo Solution - Double Blind | Testosterone Solution - Double Blind | Testosterone Solution - OLE
Serious Adverse Events (participants affected / at risk) | 8/356 | 4/354 | 24/558
Other Adverse Events (participants affected / at risk) | 143/356 | 148/354 | 252/558
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Solution - Double Blind (N=356) | Testosterone Solution - Double Blind (N=354) | Testosterone Solution - OLE (N=558)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Septic embolus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Solution - Double Blind (N=356) | Testosterone Solution - Double Blind (N=354) | Testosterone Solution - OLE (N=558)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 5 (5)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Gingival cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary duct obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Application site acne (General disorders) | 0 (0) | 0 (0) | 1 (1)
Application site dryness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site eczema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 3 (3) | 1 (1) | 4 (4)
Application site irritation (General disorders) | 0 (0) | 2 (2) | 3 (3)
Application site pain (General disorders) | 7 (7) | 6 (6) | 2 (2)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 1 (1)
Application site rash (General disorders) | 0 (0) | 0 (0) | 4 (4)
Application site reaction (General disorders) | 1 (1) | 0 (0) | 1 (1)
Application site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst rupture (General disorders) | 0 (0) | 1 (1) | 0 (0)
Effusion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4) | 2 (2)
Haemorrhagic cyst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 2 (2)
Local swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 3 (3)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Therapeutic response unexpected (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Application site pustules (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 3 (4) | 1 (1) | 7 (7)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Chest wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 6 (6) | 0 (0) | 0 (0)
Erythema induratum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 5 (5)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 3 (3) | 10 (10)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasal vestibulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (11) | 8 (8) | 19 (21)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3) | 5 (6)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 8 (9) | 19 (20)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood follicle stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Blood insulin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood luteinising hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Blood testosterone increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 2 (2) | 0 (0)
Electrocardiogram p wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Haematocrit increased (Investigations) | 2 (2) | 9 (9) | 28 (28)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
High density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Lymph node palpable (Investigations) | 0 (0) | 0 (0) | 1 (1)
Mean cell volume increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prostatic specific antigen (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prostatic specific antigen abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 2 (2) | 4 (4) | 6 (6)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 4 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Vitamin b complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8) | 6 (7)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 16 (16)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 4 (5) | 6 (7) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 4 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 3 (3) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep phase rhythm disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Writer's cramp (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (4)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 6 (6)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (3)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Libido increased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Middle insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Personality disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Premature ejaculation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (3)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 3 (3)
Genital paraesthesia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Nipple disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 1 (1)
Painful erection (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Spermatic cord pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular atrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (5)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 10 (11)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 4 (4) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (5) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Alcohol use (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Sexual activity increased (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Substance use (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Corneal transplant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
High frequency ablation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 2 (2)
Orthodontic procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Posterior lens capsulotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Suture insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Vasectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 4 (4) | 4 (4)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days